CLINICAL TRIAL: NCT06401252
Title: Effects Of Mindfulness-Based Intervention on Psychological Health Among Jordanian Nurses Taking Care Patients With Covid-19
Brief Title: Mindfulness for Nurses' Psychological Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hossam Najjem Alhawatmeh, Associate professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022 / 147 / 32
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Psychological Well-Being; Nurse's Role
Keywords: Mindfulness-based intervention, Stress, Depression, Anxiety, Nurses, COVID-19.
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders; COVID-19

STUDY DESIGN:
Intervention Model Description: two-group, randomized controlled design
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor) The data were collected by a research assistant with good nursing experiences who were not involved in any other parts of the study.
  Also, the participants were randomly assigned equally to the study groups using a computerized random numbers procedure carried out by a research assistant who was not involved in any other parts of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurses receiving Mhealth-based mindfulness-based intervention (Experimental): The experimental group received five individuals 30-minute sessions of MBI for five weeks in a private and quiet room at the hospital, according to Smith's (2005) recommendation. The study intervention was an audio based MBI sent to them by the WhatsApp application. It is a free, self-paced program developed by an experienced, certified mindfulness practitioner based on the Smith's (2005) protocol to guarantee greater adherence and consistent delivery of MBI. The audio recording of the MBI was evaluated and validated for the clarity of voice and the MBI content by two psychologists who are experts in MBI.
  Interventions: Behavioral: Mindfulness-based intervention
- Control group receiving traditional care (No Intervention): Participants in the control group were not asked to do anything during the study, except their traditional practices. However, the MBI was provided to them after the study.

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — • The mindful mediators are asked to act as neutral observers who view the world as it is, without reactions, judgments, and evaluations. They quietly attend to, note, and let go of every internal external stimulus such as thought, feeing, sensation, sound, idea that enters awareness. They do not try to think about, push away, and do anything with these stimuli experienced and do not have to figure out the connections between each 19 stimuli. They simply let each stimulus come and go and wait for the next stimulus. They do not have to be concerned about distractions. Each time they are distracted, they note it as yet another passing stimulus (Ah, a distraction… how interesting")
  Arms: Nurses receiving Mhealth-based mindfulness-based intervention

SUMMARY:
Background: Nurses who worked with patients with COVID-19 in hospitals have experienced several threatening and challenging situations, negatively affecting psychological health. M-health-based mindfulness-based interventions were found to improve psychological health in various populations.

Aim: The purpose of this study is to assess the effectiveness of a m-Health-based mindfulness-based intervention on anxiety, depression, stress among Jordanian registered nurses taking care of COVID-19 patients.

Methodology: The study was conducted using a pretest post-test randomized controlled design. One hundred and two nurses were recruited from a Jordanian Hospital and randomly distributed into experimental group (n=51) and control group (n= 51). The study data were collected using a self-report questionnaire working in the King Abdullah University hospital at baseline and at the end of intervention. For five weeks, the experimental group had five individual 30-minute MBI sessions. An audio-based MBI that was given to them via the WhatsApp served as the research intervention. A self-report questionnaire was used to collect the study data as follows: 1) demographic characteristics and 2) Mindful Attention Awareness, and 3) Scale the Depression, Anxiety, and Stress Scale (DASS-21). The study outcomes were measured at baseline and at the end of the intervention. Data were analyzed using the Statistical Package for Social Science (SPSS), Version 26.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19), first reported in Wuhan China, has been described as the first pandemic contributed to a coronavirus that has drawn intense attention worldwide. Up to April 11th, 2020, at least 381 diagnosed cases and 7 deaths have been reported in Jordan (Jordanian Health Ministry, 2020). Facing this critical situation, nurses are struggling on the front line to manage patients with COVID-19, placing them at risk of contracting the infectious disease (World Health Organization (WHO), 2020).

Like other countries, health care providers in Jordan account for a significant share of their Covid-19 cases (Jordanian Health Ministry, 2020). Although Jordanian government has undertaken much efforts to provide healthcare providers with personal protective equipment and immunization to avoid contracting the disease, their psychological well-being, like in other countries, have been disregarded (Duan, & Zhu, 2020; Huffington & Williams, 2020). A combination of long shifts, understaffing, overwhelming workload, and lack of sleep may all contribute to stress and mental burden of these healthcare providers, compromising immune systems and make them more vulnerable to the infectious disease (Chen, et al., 2020; WHO, 2020). The psychological effect experienced by nurses during the COVID-19 pandemic was evident in the literature. Anxiety, stress, and depression were commonly reported by nurses during the COVID-19 pandemics (Pratiwi, et al., 2023) Nurses' health in hospital settings is the most important consideration for providing excellent patient care. To achieve the optimal outcomes for the patients and their families, it is required that nurses to be kept at the highest level of psychological health. Therefore, officials and those in charge of health institutions must find appropriate solutions to help nurses to cope with mental health problems. A possible solution to nurses' mental health problems may rest in promoting medical interventions such as mind- body interventions (Goyal, et al., 2014).

Mindfulness-based intervention (MBI) is one of the most popular mind-body therapy methods used recently in psychotherapy, which is strongly associated with promotion physical and psychological well-being, it is an effective method for reducing stress and improving health (Bartlett, et al., 2021). Pascoe et al. (2017) imagined it as a combination of five main components: act with awareness, internal observation and external experiences, being non-judgmental, description and labeling and not reacting to thoughts and feelings. Theoretically, practicing MBI develops mindfulness trait, and then relaxes the body and mind and helps reduce the response or reactivity to stressful situation, traumatic events and challenging experiences (Hofmann & Gómez, 2017). Many researchers have pointed to the effectiveness of in-person mindfulness training programs in reducing nurses' stress, anxiety, and depression in general health settings (Ghawadra, et al. 2020; Green & Kinchen, 2021; Lomas, et al. 2019; Ramachandran, et al. 2022; Sulosaari, et al. 2022).

Mindfulness-based intervention (MBI) as a Mind-body therapy, recently increasing its popularity in Jordan, are easily accessible, easy to learn and inexpensive (Yanyu, et al., 2020). For easily accessible and nonphysical contact training mode, they can be delivered quite efficiently by easy-to-carry electronic devices to healthcare providers (Kubo, et al., 2019; Wiseman, et al., 2018). M-Health-based intervention is an innovative approach of treatment delivery using mobile technologies such as cell phones (Kubo, et al., 2019). Mobile phones are widely used in Jordan, with the most Jordanians (95%) having a smart phone (Gazal, 2020). The widespread use of smart phones highlights their potential to deliver cost-effective mind-body therapies that can be easily integrated into the lives of busy healthcare providers who are unable to attend regular in-person training sessions (Kubo, et al., 2019; Wiseman, et al., 2018). It also provides a feasible and effective therapeutic way to optimize physical distancing during pandemics, which contributes to decrease the transmission of infection (Tukur et al., 2023) Although a wide array of research has been conducted examining the relationship between MBI and psychological health problems in different populations (McGee, et al., 2023), this study came as first study-to the best of research knowledge- to examine the effectiveness of m-health-based MBI on stress, anxiety, and depression among nurses taking care patients with COVID-19. Investigating the effects of MBI on psychological health in such nurses may contribute to the development of evidence-based methods and guidelines for enhancing the mental well-being of them during this unprecedented epidemic and may also enhance humanity's ability to respond to other emerging pandemics.

Design This was an experimental study using pretest post-test randomized controlled design.

3.2 Sample Nurses taking care patients with COVID-19 in the King Abdullah University hospital (KAUH) who were aged at least 21 years old, had smart phones, and were able to read and write in English, were included. KAUH designated by the Jordanian Ministry of Health as the main COVID-19 testing and isolation center in the country's north. Participants who had psychological therapies or medications were excluded.

Using G* Power software 3.1 (Faul et al., 2007), independent t-test, an alpha of 0.05, a power of 0.8, and a moderate effect size of 0.5, a sample size of 102 was generated.

The sample was distributed randomly into the experimental group (n=61) and the control group (n= 61).

3.4 Intervention The experimental group received five individuals 30-minute sessions of MBI for five weeks in a private and quiet room at the hospital, according to Smith's (2005) recommendation. The study intervention was an audio based MBI sent to them by the WhatsApp application. It is a free, self-paced program developed by an experienced, certified mindfulness practitioner based on the Smith's (2005) protocol to guarantee greater adherence and consistent delivery of MBI. The audio recording of the MBI was evaluated and validated for the clarity of voice and the MBI content by two psychologists who are experts in MBI.

However, an instructional session, other than the five weekly sessions mentioned above, was first conducted by the certified mindfulness practitioner to explain the rationale and procedures of MBI including a demonstration of the entire MBI protocol for the participants in the experimental group. This practitioner was also present during the delivery of the five MBI sessions in the hospital to confirm and facilitate the administration of the MBI sessions and answer any participants' questions. In addition, the experimental groups' participants were encouraged to practice the intervention daily at home, but home-based practice was not mandatory. Through the WhatsApp group, daily reminders were sent to the participants in the experimental group to encourage them to practice at home. Diaries was used by the experimental group's participants to document the daily home-based practices. The participants in the experimental groups were encouraged not to share any information regarding the MBI with anyone during the study.

The theory-based program includes the ABC standardized versions of MBI (Smith, 2005), described as follows:

* The mindful mediators are asked to act as neutral observers who view the world as it is, without reactions, judgments, and evaluations. They quietly attend to, note, and let go of every internal external stimulus such as thought, feeing, sensation, sound, idea that enters awareness. They do not try to think about, push away, and do anything with these stimuli experienced and do not have to figure out the connections between each 19 stimuli. They simply let each stimulus come and go and wait for the next stimulus. They do not have to be concerned about distractions. Each time they are distracted, they note it as yet another passing stimulus (Ah, a distraction… how interesting") (Smith, 2005).
* Participants in the control group were not asked to do anything during the study, except their traditional practices. However, the MBI was provided to them after the study.

3.5 Measurements The study data were collected using a self-report questionnaire at baseline and at the end of intervention. The participants were asked to complete the study self-report questionnaire, including three parts, as follows: 1) demographic characteristics, and 2) The Depression, Anxiety, and Stress Scale (DASS-21), and 3) Mindful attention Awareness Scale 3.5.1 Demographic and Health Characteristics The demographic and health characteristics included sex, marital status, religion, department, educational level, nursing experience (years), having chronic diseases, age, weight, monthly income, general health status, nutritional status, sleeping status.

3.5.2 The Depression, Anxiety, and Stress Scale (DASS-21) The Arabic DASS was used to measure depression, anxiety and stress in the current study (Lovibond & Lovibond, 1995). The DASS-21 is a set of three self-report scales designed to measure the negative emotional states of depression, anxiety and stress. Each of the three DASS subscales contains 7 items. Subjects were asked to use 4-point severity/frequency scales to rate the extent to which they had experienced each state. Scores for Depression, Anxiety and Stress were calculated by summing the scores for the relevant items, and then multiplying the summed scores by 2. The score range of each subscale is between 0.0 to 42. Higher scores of the three subscales indicate higher levels of those emotional states. The DASS has shown acceptable levels of validity and reliability in clinical and healthy populations (Lovibond & Lovibond, 1995). The reliability and validity of Arabic version of DASS demonstrated acceptable reliability and validity of this tool (Alharbi et al. 2023). In Jordanian nursing students, the Cronbach's alphas for the stress, anxiety, and depression subscales were .73, .82, and .80 respectively (Alhawatmeh et al., 2022).

3.5.3. the Mindful Attention Awareness Scale (MAAS) was used to measure trait mindfulness. The MAAS is one-dimensional and comprises 15 items measured on a six-point Likert-type scale ranging from 1 (almost always) to 6 (almost never). The score range is between 15 and 90, with higher scores indicating higher levels of trait mindfulness. The Arabic MAAS has been shown to have excellent internal consistency and convergent validity among an Arab population.

3.6 Data collection and Ethical consideration After getting the IRB approval, the hospital administrators were contacted by the study researchers to obtain approval for conducting the study. After approval, the nurses were contacted in person by one of the study researchers to explain the study purpose and procedure. If they agreed to participate, the nurses were asked to sign the consent form. After that, a study researcher who was not involved in the recruitment process and patient assessment randomly assigned the participants to the intervention group or the control group, using a simple 1:1 computer-generated sequence. Then, the schedule of practicing the MBI as the protocol described above was given for the participants in the experimental group, which was built based on their work schedule.

The study measurements were taken at the hospital by one of the study researchers (nurses) at baseline and at the end of the intervention. Also, all study measurements in the intervention and control groups were undertaken in the same conditions (i.e., same room temperature and environment) by a well-trained nurse who has a master's degree in nursing science.

3.7 Statistical Analysis Data were analyzed using the Statistical Package for Social Science (SPSS), Version 26. Descriptive statistics were used to describe the study participants as appropriate. For instance, frequency and percentage were used to describe the categorical variables, while mean and standard deviation (SD) were used to describe the continuous variables. Also, the baseline statistical equivalence between the study groups on the dependent and sociodemographic variables was evaluated using independent t-tests. Dependent t-tests were used to examine if there were statistically significant changes between the pretest and posttest in each study group. Finally, independent t-tests were used to examine if there was a statistically significant difference between the experimental and control group at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Nurses taking care patients with COVID-19 in the King Abdullah University hospital (KAUH) who were aged at least 21 years old
* had smart phones

Exclusion Criteria:

* Participants who had psychological therapies or medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Depression, anxiety, and Stress Scale (DASS-21) | 6 weeks
  The Arabic DASS was used to measure depression, anxiety and stress in the current study (Lovibond & Lovibond, 1995). The DASS-21 is a set of three self-report scales designed to measure the negative emotional states of depression, anxiety and stress. Each of the three DASS subscales contains 7 items. Subjects were asked to use 4-point severity/frequency scales to rate the extent to which they had experienced each state. The score range of each subscale is between 0.0 to 42. Higher scores of the three subscales indicate higher levels of those emotional states. The DASS has shown acceptable levels of validity and reliability in clinical and healthy populations (Lovibond & Lovibond, 1995).
Mindful Attention awareness Scale | 6 weeks
  Mindful Attention Awareness Scale (MAAS-15) was used to assess dispositional mindfulness (Brown & Ryan, 2003).
  The Arabic version of MASS-15 is a valid and reliable scale (Rayan & Ahmad, 2018). It is one-dimensional scale including 15 items measured on a six-point likert type scale, ranging from 1 (almost always) to 6 (almost never). The score range is between 15 and 90, with higher score indicting higher levels of mindfulness. The scale has shown strong psychometric properties when validated in college students. It showed single-factor construct in MAAS structure and a Chronbach's alpha of 0.82 in university sample (Brown & Ryan, 2003).

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University of Science and Technology, Irbid, None Selected, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhawatmeh H, Albataineh R, Abuhammad S. Differential effects of guided imagery and progressive muscle relaxation on physical and emotional symptoms in nursing students taking initial clinical training: A randomized clinical trial. Heliyon. 2022 Oct 19;8(10):e11147. doi: 10.1016/j.heliyon.2022.e11147. eCollection 2022 Oct. PMID 36311359
- [Background] Alharbi, F. S., Gangwani, S., Alsubaie, B. A., Osman, M., Alotaibi, F. S., Alsamman, D. D., & Mahfouz, T. A. O. (2023). Depression, Anxiety, and Stress among Adults in Saudi Arabia. Resmilitaris, 13(3), 1664-1672.
- [Background] Al Ozairi A, Alsaeed D, Al-Ozairi E, Irshad M, Crane RS, Almoula A. Effectiveness of virtual mindfulness-based interventions on perceived anxiety and depression of physicians during the COVID-19 pandemic: A pre-post experimental study. Front Psychiatry. 2023 Jan 9;13:1089147. doi: 10.3389/fpsyt.2022.1089147. eCollection 2022. PMID 36699484
- [Background] Bartlett L, Buscot MJ, Bindoff A, Chambers R, Hassed C. Mindfulness Is Associated With Lower Stress and Higher Work Engagement in a Large Sample of MOOC Participants. Front Psychol. 2021 Sep 10;12:724126. doi: 10.3389/fpsyg.2021.724126. eCollection 2021. PMID 34566805
- [Background] Chen Q, Liang M, Li Y, Guo J, Fei D, Wang L, He L, Sheng C, Cai Y, Li X, Wang J, Zhang Z. Mental health care for medical staff in China during the COVID-19 outbreak. Lancet Psychiatry. 2020 Apr;7(4):e15-e16. doi: 10.1016/S2215-0366(20)30078-X. Epub 2020 Feb 19. No abstract available. PMID 32085839
- [Background] Duan L, Zhu G. Psychological interventions for people affected by the COVID-19 epidemic. Lancet Psychiatry. 2020 Apr;7(4):300-302. doi: 10.1016/S2215-0366(20)30073-0. Epub 2020 Feb 19. No abstract available. PMID 32085840
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Gazal, M. (2020). 95% of Jordanians own mobiles; 47% use the Internet. The Jordan Times. Retrieved from: http://www.jordantimes.com/news/local/95-jordanians-own-mobiles-47-use-internet
- [Background] Ghawadra SF, Lim Abdullah K, Choo WY, Danaee M, Phang CK. The effect of mindfulness-based training on stress, anxiety, depression and job satisfaction among ward nurses: A randomized control trial. J Nurs Manag. 2020 Jul;28(5):1088-1097. doi: 10.1111/jonm.13049. Epub 2020 Jun 24. PMID 32432795
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Green AA, Kinchen EV. The Effects of Mindfulness Meditation on Stress and Burnout in Nurses. J Holist Nurs. 2021 Dec;39(4):356-368. doi: 10.1177/08980101211015818. Epub 2021 May 17. PMID 33998935
- [Background] Hofmann SG, Gomez AF. Mindfulness-Based Interventions for Anxiety and Depression. Psychiatr Clin North Am. 2017 Dec;40(4):739-749. doi: 10.1016/j.psc.2017.08.008. Epub 2017 Sep 18. PMID 29080597
- [Background] Huffington, A & Williams, M. (2020). Combating coronavirus starts with keeping health workers well (commentary). Fortune. Retrieved from: https://fortune.com/2020/03/11/coronavirus-health-care-workers-well-being/
- [Background] Jordanian Health Ministry. (2020). Coronavirus. Retrieved from: https://corona.moh.gov.jo/ar
- [Background] Kubo A, Kurtovich E, McGinnis M, Aghaee S, Altschuler A, Quesenberry C Jr, Kolevska T, Avins AL. A Randomized Controlled Trial of mHealth Mindfulness Intervention for Cancer Patients and Informal Cancer Caregivers: A Feasibility Study Within an Integrated Health Care Delivery System. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419850634. doi: 10.1177/1534735419850634. PMID 31092044
- [Background] Kwok, S. Y., Gu, M., & Kit, K. T. (2016). Positive psychology intervention to alleviate child depression and increase life satisfaction: A randomized clinical trial. Research on social work practice, 26(4), 350-361. https://doi.org/10.1177/10497315166297
- [Background] Lan, H. K., Subramanian, P., Rahmat, N., & Kar, P. C. (2014). The effects of mindfulness training program on reducing stress and promoting well-being among nurses in critical care units. Australian Journal of Advanced Nursing, 31(3), 22-31.
- [Background] Lomas, T., Medina, J. C., Ivtzan, I., Rupprecht, S., & Eiroa-Orosa, F. J. (2019). A systematic review and meta-analysis of the impact of mindfulness-based interventions on the well-being of healthcare professionals. Mindfulness, 10(7), 1193-1216. https://doi.org/10.1007/s12671-018-1062-5
- [Background] Lovibond, S. H., & P.F. Lovibond, P. F. Manual for the Depression Anxiety Stress Scales. Psychology Foundation, Sydney, 1995.
- [Background] McGee, A. B., Scott, S. R., Manczak, E. M., & Watamura, S. E. (2023). Associations between the Psychophysiological Impacts of Teacher Occupational Stress and Stress Biomarkers: A Systematic Review. Psychoneuroimmunology Journal, art246145. DOI:10.32371/pnij/246145
- [Background] Pascoe MC, Thompson DR, Jenkins ZM, Ski CF. Mindfulness mediates the physiological markers of stress: Systematic review and meta-analysis. J Psychiatr Res. 2017 Dec;95:156-178. doi: 10.1016/j.jpsychires.2017.08.004. Epub 2017 Aug 23. PMID 28863392
- [Background] Pratiwi, I. N., Nihayati, H. E., Santus, R., Ramoo, V., & Nursalam, N. (2023). Psychological impacts of the COVID-19 pandemic on nurses and coping strategies: a systematic review. Journal of Public Health and Emergency, 7, 1-15. doi: 10.21037/jphe-22-57
- [Background] Ramachandran HJ, Bin Mahmud MS, Rajendran P, Jiang Y, Cheng L, Wang W. Effectiveness of mindfulness-based interventions on psychological well-being, burnout and post-traumatic stress disorder among nurses: A systematic review and meta-analysis. J Clin Nurs. 2023 Jun;32(11-12):2323-2338. doi: 10.1111/jocn.16265. Epub 2022 Feb 20. PMID 35187740
- [Background] Sari YP, Hsu YY, Nguyen TTB. The Effects of a Mindfulness-Based Intervention on Mental Health Outcomes in Pregnant Woman: A Systematic Review and Meta-Analysis. J Nurs Res. 2023 Dec 1;31(6):e306. doi: 10.1097/jnr.0000000000000586. PMID 38036493
- [Background] Smith, J. C. (2005). Relaxation, meditation, & mindfulness: A mental health practitioner's guide to new and traditional approaches. Springer Publishing Company.
- [Background] Spinelli C, Wisener M, Khoury B. Mindfulness training for healthcare professionals and trainees: A meta-analysis of randomized controlled trials. J Psychosom Res. 2019 May;120:29-38. doi: 10.1016/j.jpsychores.2019.03.003. Epub 2019 Mar 5. PMID 30929705
- [Background] Sulosaari V, Unal E, Cinar FI. The effectiveness of mindfulness-based interventions on the psychological well-being of nurses: A systematic review. Appl Nurs Res. 2022 Apr;64:151565. doi: 10.1016/j.apnr.2022.151565. Epub 2022 Jan 15. PMID 35307128
- [Background] Tukur M, Saad G, AlShagathrh FM, Househ M, Agus M. Telehealth interventions during COVID-19 pandemic: a scoping review of applications, challenges, privacy and security issues. BMJ Health Care Inform. 2023 Aug;30(1):e100676. doi: 10.1136/bmjhci-2022-100676. PMID 37541739
- [Background] van der Riet P, Levett-Jones T, Aquino-Russell C. The effectiveness of mindfulness meditation for nurses and nursing students: An integrated literature review. Nurse Educ Today. 2018 Jun;65:201-211. doi: 10.1016/j.nedt.2018.03.018. Epub 2018 Mar 24. PMID 29602138
- [Background] Lehto RH, Heeter C, Allbritton M, Wiseman M. Hospice and Palliative Care Provider Experiences With Meditation Using Mobile Applications. Oncol Nurs Forum. 2018 May 1;45(3):380-388. doi: 10.1188/18.ONF.380-388. PMID 29683121
- [Background] Yanyu, J., Xi, Y., Huiqi, T., Bangjiang, F., Bin, L., Yabin, G., … Lijun, J. (2020). Meditation-based interventions might be helpful for coping with the Coronavirus disease 2019(COVID-19). https://doi.org/10.31219/osf.io/f3xzq
- [Background] Young, N. (2021). What are the social determinants of good mental and physical health? Nursing Times [online], 117(10), 21-24.
- [Derived] Alhawatmeh H, Abusaif L, Alharrasi M, AbuAlrub RF, Hamaideh SH. Holistic Healing Through Mindfulness: An Experimental Study Addressing Psychological Challenges Among Nurses Caring for Patients With COVID-19. J Holist Nurs. 2025 Mar 17:8980101251323021. doi: 10.1177/08980101251323021. Online ahead of print. PMID 40095566